CLINICAL TRIAL: NCT02935712
Title: A Phase I, Randomized, Single-Blind, Placebo Controlled Study to Assess the Safety, Tolerability and Pharmacodynamics Of AZD8601 After Single Dose Administration to Male Patients With Type II Diabetes Mellitus (T2DM)
Brief Title: Assessment of the Safety, Tolerability and Pharmacodynamics After Administration of One Dose of AZD8601 to Male Patients With Type II Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry); Spandauer Damm 130 (Unknown); 14050 (Unknown); Berlin, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D9150C00001; 2016-002316-40 (EudraCT Number)
Record Dates: First submitted 2016-08-18; First posted 2016-10-17 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Male Subjects With Type II Diabetes (T2DM)
Keywords: Safety; Tolerability; AZD8601; Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sagittal Abdominal Diameter; Placebo Effect

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Three cohorts with 9 subjects and each cohort received 2 treatments (AZD8601+Placebo/ Placebo+Placebo)
  Interventions: Drug: AZD8601+Placebo (SAD); Drug: Placebo+Placebo
- Part B (Experimental): Subjects received 2 treatments (AZD8601+Placebo)
  Interventions: Drug: AZD8601+Placebo

INTERVENTIONS:
Drug: AZD8601+Placebo (SAD) — Six subjects are randomized to receive one treatment of AZD8601 and one treatment of Placebo.
  Single ascending dose (SAD) with a sequential cohort design and three dose levels of AZD8601 are planned to be investigated. Subjects will receive 0.004 mg per injection of AZD8601/placebo with a total proposed dose of 0.024 mg.
  Arms: Part A
Drug: AZD8601+Placebo — Subjects will receive dose with sufficient vascular endothelial growth factor (VEGF)-A protein production and a good safety profile as determined in Part A and the total dose per patient will not exceed the maximum dose given in Part A.
  Arms: Part B
Drug: Placebo+Placebo — Subjects are randomized to receive 2 placebo treatments.
  Arms: Part A

SUMMARY:
This study will be a phase I, first time in human (FiH), randomized, single-blind, placebo-controlled, SAD study in male patients with T2DM, performed at a single study center. The study will consist of 2 parts, (A and B) up to 60 male patients with T2DM aged 18 to 65 years will be included

DETAILED DESCRIPTION:
Part A will assess the safety and tolerability of SAD of intradermal (ID) injection of AZD8601 (modified VEGF-A RNA) and Part B will evaluate the pharmacodynamic effects of ID injection of AZD8601 in forearm skin. AZD8601 is a VEGF-A modified RNA under development as a novel modality for local production of human VEGF-A protein and is developed for the treatment of diabetic patients with ulcers. Each patient in Part A will be involved in the study for 7 to 8 weeks. Each patient in Part B will be involved in the study for 5 to 6 weeks.

Safety and tolerability variables includes Adverse events (AEs), Vital signs (BP, pulse), ECG, Hematology, Clinical chemistry, Urinalysis.

The study will include patients with T2DM that are on stable doses of 1 to 2 anti-diabetic medications. The T2DM patients may also be on medications for comorbidities such as hypertension, dyslipidemia, hyperuricemia, thyroid disorders, benign prostate hyperplasia etc. (e.g. diuretics, statins, allopurinol, thyroxin), but must be healthy otherwise.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Male patients with mild T2DM aged 18 to 65 years with suitable veins for cannulation or repeated venipuncture.
3. Have a body mass index (BMI) between 20 and 35 kg/m2 inclusive and weigh at least 50 kg.
4. Able to understand, read and speak the German language.
5. T2DM diagnosis for at least 1 year at the time of the screening visit.
6. T2DM treated with diet and exercise alone or with up to 2 oral anti-diabetic drugs.
7. Have stable glycemic control indicated by no changed treatment within 3 months prior to enrolment.
8. Hemoglobin A1c less than 10.5% at screening (HbA1c value according to international Diabetes Control and Complications Trial standard).
9. Fasting plasma glucose ≤ 11.0 mmol/L at screening.
10. Provision of signed, written and dated informed consent for optional genetic/biomarker research.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study.
2. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the before Day -1
3. Any clinically significant abnormalities in clinical chemistry, hematology or urinalysis results at screening and check-in, as judged by the PI.

   The following strict criteria will apply at the time of screening and on Day -1:
   * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) > 2 times the upper limit of the normal laboratory range
   * Hemoglobin < 11 g/dL and/or neutrophils < 1500/mm3 and/or platelets < 100 000/mm3
   * Creatinine > 1.2 x upper limit of normal (ULN)
4. Uncontrolled or inadequately controlled hypertension at the time of screening and/or on Day -1 with a resting systolic or diastolic BP > 150 mmHg or > 95 mmHg, respectively. Patients with heart rate < 50 bpm at screening and on Day -1 will be excluded.
5. Any clinically significant abnormalities on 12-lead ECG at screening as judged by the PI.
6. Any patient with QT interval corrected for heart rate using Fridericia's formula (QTcF) > 450 ms at screening should be excluded.
7. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), anti-hepatitis B core (HBc) antibody, hepatitis C antibody and human immunodeficiency virus (HIV) antibody.
8. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of Day -1 of this study. The period of exclusion begins 3 months after the final dose from a previous study or 1 month after the last visit, whichever is longer. 9. Plasma donation within 1 month of screening or any blood donation/loss more than 400 mL during the 3 months prior to screening.

10. Current smokers or those who have smoked or used nicotine products within the previous 1 year cotinine below the cut-off of the local laboratory).

11. Positive screen for drugs of abuse, cotinine or alcohol at screening or admission to the study center.

12. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the PI.

13. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/ acetaminophen), herbal remedies, mega-dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to admission or longer if the medication has a long half-life.

Patients with T2DM can be on 1 to 2 anti-diabetic medications but need the medication to be on stable doses for at least 3 months. Patients with T2DM can also be on medications for comorbidities such as hypertension, dyslipidemia, hyperuricemia, thyroid disorders, benign prostate hyperplasia etc. (e.g. diuretics, statins, allopurinol, thyroxin) but need to be on a stable dose for at least 3 months.

14. Involvement of any AstraZeneca or study site employee or their close relatives.

15. Judgment by the PI that the patient should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.

16. Vulnerable patients, e.g., kept in detention, protected adults under guardianship, trusteeship or committed to an institution by governmental or juridical order.

17. Reports a significant history of allergy to soaps, lotions, emollients, ointments, creams, cosmetics, adhesives or latex.

18. Reports a history of significant skin conditions or disorders, for example, psoriasis, atopic dermatitis, etc.

19. Reports a history of significant dermatologic cancers, for example, melanoma or squamous cell carcinoma. Basal cell carcinomas that were superficial or successfully removed or treated, and do not involve the investigative site are acceptable.

20. Presence of forearm tattoo(s). 21. History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening.

22. History of myocardial infarction, stroke, or heart failure requiring hospitalization within 6 months prior to the time of screening, history or presence of clinically significant diabetic retinopathy, history or presence of macular edema likely to require LASER treatment within the study period.

23. Uncontrolled cardiovascular, hepatic, neurological or endocrine disease. 24. Use of insulin, glitazones, warfarin and amiodarone within 3 months before enrolment and use of potent CYP450 inhibitors, e.g., ketoconazole and macrolide antibiotics within 14 days before screening.

25. Use of anabolic steroids and systemic treatment with glucocorticoids within 3 months before screening.

26. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea, chocolate), as judged by the PI 27. Patients who cannot communicate reliably with the PI. In addition, any of the following is regarded as a criterion for exclusion from the genetic research: 28. Previous bone marrow transplant 29. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Safety of AZD8601 by assessing summary of adverse events (Part A) | Part A: From screening (Day -28) up to Day 29
  To evaluate the safety by assessing the adverse event after administration of a single dose of AZD8601 to male subjects with T2DM (Part A).
Safety of AZD8601 by assessing number of subjects with clinically significant blood pressure (Part A) | Part A: Day 1 to Day 8
  To evaluate the safety by assessing the number of subjects with clinically significant blood pressure after administration of single dose of AZD8601 to male subjects with T2DM (Part A).
Safety of AZD8601 by assessing number of subjects with Clinically significant pulse (Part A) | Part A: Day 1 to Day 8
  To evaluate the safety by assessing the number of subjects with clinically significant pulse after administration of single dose of AZD8601 to male subjects with T2DM (Part A).
Safety of AZD8601 by assessing number of subjects with Clinically significant 12-lead electrocardiograms (ECGs) (Part A) | Part A: Day 1 to Day 8
  To evaluate the safety by assessing the number of subjects with clinically significant ECGs after administration of single dose of AZD8601 to male subjects with T2DM (Part A).
Safety of AZD8601 by assessing number of subjects with clinically significant hematology parameters (Part A) | Part A: Day 1 to Day 8
  To evaluate the safety by assessing the number of subjects with clinically significant hematology parameters after administration of single dose of AZD8601 to male subjects with T2DM (Part A).
Safety of AZD8601 by assessing number of subjects with clinically significant clinical chemistry laboratory results (Part A) | Part A: Day 1 to Day 8
  To evaluate the safety by assessing the number of subjects with clinically significant clinical chemistry laboratory results after administration of single dose of AZD8601 to male subjects with T2DM (Part A).
Safety of AZD8601 by assessing number of subjects with clinically significant urinalysis (Part A) | Part A: Day 1 to Day 8
  To evaluate the safety by assessing the number of subjects with clinically significant urinalysis after administration of single dose of AZD8601 to male subjects with T2DM (Part A).
Safety of AZD8601 by assessing summary of adverse events (Part B) | Part B: From screening up to Day 15
  To evaluate the safety by assessing the adverse event after administration of a single dose of AZD8601 to male subjects with T2DM (Part B).
Safety of AZD8601 by assessing number of subjects with clinically significant blood pressure (Part B) | Part B: Day 1 to Day 2
  To evaluate the safety by assessing the number of subjects with clinically significant blood pressure after administration of single dose of AZD8601 to male subjects with T2DM (Part B).
Safety of AZD8601 by assessing number of subjects with Clinically significant pulse (Part B) | Part B: Day 1 to Day 2
  To evaluate the safety by assessing the number of subjects with clinically significant pulse after administration of single dose of AZD8601 to male subjects with T2DM (Part B).
Safety of AZD8601 by assessing number of subjects with Clinically significant 12-lead electrocardiograms (ECGs) (Part B) | Part B: Day 1 to Day 2
  To evaluate the safety by assessing the number of subjects with clinically significant ECGs after administration of single dose of AZD8601 to male subjects with T2DM (Part B).
Safety of AZD8601 by assessing number of subjects with clinically significant hematology parameters (Part B) | Part B: Day 1 to Day 2
  To evaluate the safety by assessing the number of subjects with clinically significant hematology parameters after administration of single dose of AZD8601 to male subjects with T2DM (Part B).
Safety of AZD8601 by assessing number of subjects with clinically significant clinical chemistry laboratory results (Part B) | Part B: Day 1 to Day 2
  To evaluate the safety by assessing the number of subjects with clinically significant clinical chemistry laboratory results after administration of single dose of AZD8601 to male subjects with T2DM (Part B).
Safety of AZD8601 by assessing number of subjects with clinically significant urinalysis (Part B) | Part B: Day 1 to Day 2
  To evaluate the safety by assessing the number of subjects with clinically significant urinalysis after administration of single dose of AZD8601 to male subjects with T2DM (Part B).

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, Dr. med., Principal Investigator — Early Phase Clinical Unit, PAREXEL International GmbH, Berlin
Locations (1):
- Research Site, Berlin, Germany